CLINICAL TRIAL: NCT05436990
Title: A Phase II Multicenter Study to Assess the Antitumor Activity of Vactosertib in Combination With Pembrolizumab in Acral and Mucosal Melanoma Patients Progressed From Prior Immune Check Point Inhibitor
Brief Title: Antitumor Activity of Vactosertib in Combination With Pembrolizumab in Acral and Mucosal Melanoma Patients Progressed From Prior Immune Check Point Inhibitor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: According to the protocol criteria, during the Phase 1 analysis, the registered participants' imaging evaluation responses did not meet the criteria, leading to an early termination
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-0713
Record Dates: First submitted 2022-06-16; First posted 2022-06-29 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Acral Melanoma; Mucosal Melanoma
MeSH Terms: interventions — pembrolizumab; vactosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vactosertib in combination with pembrolizumab (Experimental): Participants will be treated for up to 35 cycles (approximately 2 years) after initiation of treatment with intravenous 200mg of pembrolizumab every 3 weeks in combination with vactosertib. Vactosertib will be given orally for 200mg, bid for 5 days (from Mon. to Fri.) per week.
  Interventions: Drug: Pembrolizumab, Vactosertib

INTERVENTIONS:
Drug: Pembrolizumab, Vactosertib — Participants will be treated for up to 35 cycles (approximately 2 years) after initiation of treatment with intravenous 200mg of pembrolizumab every 3 weeks in combination with vactosertib. Vactosertib will be given orally for 200mg, bid for 5 days (from Mon. to Fri.) per week.

SUMMARY:
This trial is a multicenter, single arm study of efficacy of vactosertib in combination with pembrolizumab in advanced acral or mucosal melanoma patients progressed prior treatment including immunotherapy or targeted therapy and chemotherapy. This trial will be conducted though Korean Cancer Study Group (KCSG). The KCSG is responsible for the project management of the trial. Patient recruitment will take at 4 institutions.

Participants will be treated for up to 35 cycles (approximately 2 years) after initiation of treatment with intravenous 200mg of pembrolizumab every 3 weeks in combination with vactosertib. Vactosertib will be given orally for 200mg, bid for 5 days (from Mon. to Fri.) per week. This study will use ORR based on RECIST 1.1 and modified RECIST 1.1 (immune related RECIST) criteria as the primary endpoint and the tumor assessment will be done every 6 weeks. Secondary endpoints are DCR, PFS, OS, and safeties. Exploratory biomarkers predictive biomarker candidates (e.g., level of PD-L1 tumor expression, EMT marker, PD-L1, TGF-β RII, and pSMAD2) in tumor tissue and ctDNA in blood will be investigated in both pre-treatment and post-treatment periods.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of acral or mucosal melanoma with stage IV or unresectable stage III diseasewill be enrolled in this study.
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention
3. Have progressed after at least one line of therapy which must include anti-PD-1 (and/or anti-CTLA4) treatment for metastatic melanoma.

   1. patients with actionable BRAF mutation must also have been treated with appropriate targeted therapy (BRAF inhibitor and/or RAF inhibitor),
   2. patient treated with chemotherapy can be enrolled
4. Participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
   2. Has demonstrated disease progression after anti-PD-1/L1 as defined by RECIST v1.1.
5. c. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb. Patients must be able to swallow tablets and absorb vactosertib.
6. Life expectancy > 3 months
7. Patients with CNS metastasis must have stable neurologic function without evidence of CNS progression within 8 weeks (i.e., patients with controlled, asymptomatic or with resected CNS metastases with no radiological evidence of disease)
8. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
9. Male participants:

A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least [120 days, corresponding to time needed to eliminate any study treatment(s) (e.g. 5 terminal half-lives for pembrolizumab and/or any active comparator/combination) plus an additional 90 days (a spermatogenesis cycle) for study treatments with evidence of genotoxicity at any dose] after the last dose of study treatment and refrain from donating sperm during this period.

Female participants:

A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days 10. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies: 4. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days (corresponding to time needed to eliminate any study treatments (pembrolizumab and vactosertib) plus 30 days (a menstruation cycle) for study treatments with risk of genotoxicity after the last dose of study treatment.

11. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

12. Have adequate organ function as defined as following. Specimens must be collected within 10 days prior to the start of study intervention.

* Absolute neutrophil count (ANC)≥1500/µL
* Platelets≥100 000/µL
* Hemoglobin≥9.0 g/dL or ≥5.6 mmol/La
* Creatinine OR Measured or calculatedb creatinine clearance(GFR can also be used in place of creatinine or CrCl)≤1.5 × ULN OR

  ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
* Total bilirubin≤1.5 ×ULN (≤3 × ULN for participants with liver metastases) OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
* AST (SGOT) and ALT (SGPT)≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
* International normalized ratio (INR) OR prothrombin time (PT), Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to [randomization/allocation] (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
3. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
4. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
6. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
7. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
8. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
10. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
11. Has an active infection requiring systemic therapy.
12. Concurrent active Hepatitis B (defined as HBsAG positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
16. Has had an allogenic tissue/solid organ transplant.
17. Patients treated with co-administration of a strong CYP3A4 inducers (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort) or inhibitors (e.g. clarithromycin, grapefruit juice, itraconazole, ketoconazole, posaconazole, telithromycin, and voriconazole)
18. Demonstrates a QTc interval >450 ms for men or >470 ms for women, or has known history of congenital QT-prolongation or Torsade de pointes (TdP).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Primary analysis is planned at approximately 6 months after the first dose of last enrolled patient, after study termination, or at study completion decided by Principal Investigator, whichever occurs first, assessed up to 6months.
  Efficacy Analysis Set includes all patients who have received at least 1 dose of the study drug, had measurable disease at baseline according to RECIST 1.1, and had at least 1 post-baseline tumor response assessment. Patients with evidence of disease progression or death before the first scheduled assessment of tumor response will be included in this Analysis Set. It will be the primary analysis set for tumor response.
  Primary efficacy endpoints will be based upon investigators' tumor assessments per RECIST 1.1 and will be summarized as follows to evaluate the preliminary anticancer activities of vactosertib and pembrolizumab combination. Overall response rate (ORR) is defined as the proportion of patients who have a partial or complete response to therapy by RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Jung, Principal Investigator — Division of Medical Oncology, Department of Internal Medicine, Yonsei cancer center, Severance Hospital, Yonsei University Healthy System
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No